CLINICAL TRIAL: NCT00588289
Title: CCG-LTFI: A Groupwide Protocol for Collecting Follow- up Data
Brief Title: Long Term Follow-Up of Patients on Children's Cancer Group Protocols- (CCG-LTF1) FOLLOW-UP DATA
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Oncology Group (Network); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 99-068; CA42764
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Pediatric Cancers; Oncology
Keywords: Pediatric Cancers; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This protocol is not an independent research study, but rather a means to aggregate Children's Cancer Group protocols that are closed to patient entry for the purpose of collecting current status information on those patients treated under those protocols.

DETAILED DESCRIPTION:
Children's Cancer Group clinical trials are conducted to improve understanding of the biology and treatment of childhood cancers. Protocols are developed by expert committees and distributed from the Group Operations Center to the member institutions. Before a protocol can be opened to patient accrual at a CCG institution, the protocol, consent form and any activation amendments are reviewed and approved by the local Institutional Review Board QRB).

Protocols remain open to patient accrual until sufficient evaluable patients have been entered to answer the study questions. During this time, the protocol and any new amendments are reviewed annually by the IRB. When the study has been closed to patient accrual it remains open solely for the purpose of collecting life status and occurrence of adverse events. The IRB must continue its annual review as long as a patient treated on the protocol is alive and follow-up data are being collected. The CCG Long Term Follow-up protocol (CCG-LTF1) is meant to allow continued collective review of all protocols that meet the following criteria: (a) It is closed to patient accrual, (b) all patients have completed treatment, and (c) there are patients who are alive and being followed. The protocols that meet these criteria will be listed as being aggregated under CCG-LTF1 such that an IRB review of CCG-LTF1 will constitute a review of that protocol.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have completed anti-cancer treatment according to a CCG protocol, or must have been declared off protocol therapy, but not off study.
* The data to be collected on the patient must include only those data that are documented in the medical record or included on the follow-up forms.

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient must have completed anti-cancer treatment according to a CCG protocol, or must have been declared off protocol therapy, but not off study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 1999-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Facilitate reporting of adverse events for those who completed treatment; To establish a mechanism for regular annual approval; Decrease the number of active protocols; Develop a framework for future studies of long-term health related outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Steinherz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Joseph Neglia, MD, MPH, Study Chair — University of Minnesota Medical Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org